CLINICAL TRIAL: NCT05890833
Title: The FBIndex to Determine the Risk of Falls and Its Translation to Assistive Gait Device Care for Patients With Neuromuscular Disorders
Brief Title: The Risk of Falls Index for Patients With Neuromuscular Disorders
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Marko Mijic, Master of Sports and Movement Therapy, LMU Klinikum
Other Study IDs: FBIndex_80336
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Inclusion Body Myositis; Myotonic Dystrophy; Facioscapulohumeral Muscular Dystrophies; Myasthenia Gravis; The Falls Efficacy Scale International; The Morse Fall Scale
MeSH Terms: conditions — Myositis, Inclusion Body; Myotonic Dystrophy; Muscular Dystrophy, Facioscapulohumeral; Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neuromuscular disorders
  Interventions: Diagnostic Test: The risk of falls

INTERVENTIONS:
Diagnostic Test: The risk of falls — Heel-Rise-Test, Chair-Rise Test, Semi-tandem stand, Trunk Rise Test, and Foot-tapping speed. Test battery two includes Timed Up and Go test, 10 Meter Walk Test, Six Minute Walk test, The Falls Efficacy Scale International FES-I, The Morse Fall Scale.

SUMMARY:
The combination of short quantitatively assessing muscular function and balance in combination with short clinical scores, can be a new valid approach to evaluate the patient risk of fall and help to create a quick checkup test to prescribe an appropriate assistive device.

The primary goal of this project is to provide a short battery of clinical assessments used to determine risk of falling for patients with neuromuscular diseases (NMD) based on correlation between clinical assessments between two groups of NMD patients and scales used to assess risk of falling for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18- and 65-year-old
* Patients with adequate cognitive and communication function to fill out the scales assessing risk of falling
* The neuromuscular disease needs to be confirmed by genetic report and/or disease deepening neurophysiological examination.

Exclusion Criteria:

- Patients which are not able to perform motoric functional assessments without assistive gait device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Following neuromuscular diseases are included in the study: inclusion body myositis, myotonic dystrophies, limb girdle and facioscapulohumeral muscular dystrophies, and myasthenia gravis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
FBIndex | 2 years
  The primary goal of this project is to provide a short battery of clinical assessments used to determine risk of falling for patients with NMDs based on correlation between clinical assessments: Heel-Rise-Test, Chair-Rise Test, Semi-tandem stand, Trunk Rise Test, and Foot-tapping speed, Timed Up and Go test, 10 Meter Walk Test and Six Minute Walk test, between two groups of NMD patients and scales: "The Falls Efficacy Scale International FES-I" and "The Morse Fall Scale" used to assess risk of falling for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Marko Mijic, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No